CLINICAL TRIAL: NCT02941510
Title: Inhaled Budesonide for Altitude Illness Prevention
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Stopped prior to enrollment per PI and DSMB decision.
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 16-2184
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Altitude Sickness
MeSH Terms: conditions — Altitude Sickness | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Budesonide (Experimental): Will participate in all study activities but will receive budesonide.
  Interventions: Drug: Budesonide
- Placebo (Placebo Comparator): Will participate in all study activities but will receive placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Budesonide — Budesonide is FDA approved for the treatment of asthma and Chronic Obstructive Pulmonary Disease (COPD). It works by reducing lung inflammation to increase oxygen uptake by the body. The researchers are examining if this medication can prevent altitude sickness.
  Arms: Budesonide
Other: Placebo — Subject(s) will participate in all study activities but will receive placebo.
  Arms: Placebo

SUMMARY:
A randomized, double-blinded study administering budesonide, a medication to reduce inflammation in the lungs, to healthy volunteers to examine effects on altitude illness prevention by spending 18 hours overnight at 14,000 ft elevation.

DETAILED DESCRIPTION:
A randomized, double-blinded study will be conducted to validate the results of previous literature on the use of budesonide in the prevention of altitude sickness. It will be conducted using healthy participants overseen by experienced wilderness medicine and altitude researchers from the Altitude Research Center at University of Colorado Denver. Participants will be recruited from the Denver community and prescreened for eligibility via phone. 100 participants, after consenting, will have baseline data and blood collected and will begin budesonide therapy 72 hours prior to being taken from Denver to Pikes Peak, where they will be observed at altitude for 18 hours. Patients will have the opportunity to withdraw consent at any time and will be monitored continuously by physician-researchers. Data collection and blood draws will be performed at specific time points and analyzed for efficacy of budesonide vs. placebo in the incidence of altitude sickness.

ELIGIBILITY:
Inclusion Criteria:

* healthy, altitude naive, 21-40 years old

Exclusion Criteria:

* smokers
* pregnancy
* hx of asthma
* current inhaled steroid use
* those with diseases or disorders known to be affected by hypoxia or the drugs used in this study such as

  * migraine or other chronic headaches,
  * sickle cell trait or disease, or
  * diabetes
* history of significant head injury or seizures
* taking any medication (over-the-counter or prescription) or herbal supplements
* a known hypersensitivity reaction to budesonide
* inability to be headache-free when consuming the amount of caffeine in two six ounce cups of coffee or less per day
* exposure to high altitude above 2000m in the previous 1 month or
* those who have been on an airline flight over six hours (Airplane cabins are pressurized to an elevation that can approximate exposure to high altitude)

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-03-06 (Actual); Study Completion 2017-03-06 (Actual)

PRIMARY OUTCOMES:
Changes in Inflammation | During 18 hours at elevation compared to baseline.
  Analysis to compare activity in pro-inflammatory pathways and activity in anti-permeability pathways, as measured by serum markers, between budesonide and placebo.
Incidence of Acute Mountain Sickness (AMS) | During 18 hours at elevation compared to baseline.
  Comparison of incidence and severity of acute mountain sickness between budesonide and placebo.
Changes in Gene regulation | During 18 hours at elevation compared to baseline.
  Comparison of gene regulation involved in acclimatization and altitude illness.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Paterson, MD, DiMM, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No